CLINICAL TRIAL: NCT00417898
Title: Phase 1 Study to Assess the Safety of 500mg of Aspirin Added to IV TPA at Standard Doses to Prevent Re-occlusion of Cerebral Vessels After Successful Reperfusion.
Brief Title: Study of Aspirin and TPA in Acute Ischemic Stroke
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATPA-HMO-CTIL
Record Dates: First submitted 2007-01-02; First posted 2007-01-04 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2007-01

CONDITIONS: Acute Ischemic Stroke
Keywords: Stroke; Cerebral Ischemia; Tissue Plasminogen Activator; Aspirin; Human; Cerebral Reperfusion
MeSH Terms: conditions — Ischemic Stroke; Stroke; Brain Ischemia | interventions — Aspirin

INTERVENTIONS:
Drug: Aspirin

SUMMARY:
This study will determine the safety of 500mg of aspirin added to IV TPA at standard doses to prevent re-occlusion of cerebral vessels after successful reperfusion. In ischemic stroke brain arteries are occluded either by an embolus originating in the heart or large vessels leading to the brain or by a process of acute thrombosis of the cerebral arteries over a ruptured atherosclerotic plaque. Rupture of the plaque exposes thrombogenic elements within the plaque and leads to accumulation and activation of platelets and induction of the clotting cascade eventually leading to acute thrombosis and occlusion of the artery. TPA is currently approved by the Food and Drug Administration to treat heart and brain problems caused by blockage of arteries. It activates plasminogen and leads to disintegration of the thrombus/embolus. It is effective only if begun within 3 to 4.5 hours of onset of the stroke because of potential deleterious side effects including life threatening symptomatic intracranial hemorrhage (sICH) when the drug is administered outside of this time window.

Reperfusion of the ischemic brain (i.e. timely opening of the occluded artery) with TPA is associated with improved outcome. However, in about 33% of patients that have successfully reperfused after TPA the artery re-occludes within the first few hours resulting in worsening neurological symptoms and worse functional outcome. This re-occlusion is speculated to result from re-thrombosis over an existing ruptured atherosclerotic plaque. This is explained by the relatively short half life of TPA leaving the exposed ruptured plaque intact which leads to re-activation of platelets and clotting factors and re-thrombosis. Thus, we hypothesize that the addition of an antiplatelet agent to TPA would result in lower rates of re-occlusion after AIS. The FDA approved TPA for patients with AIS but discouraged the concomitant use of anti-platelet or anti-thrombotic drugs for the first 24hours after administration of TPA because of concerns that such therapy may result in increased rates of intracerebral hemorrhage. Aspirin is a well known platelet anti-aggregant that works by inhibition of cycloxygenase 1 and reduction in thromboxane A levels. It has a rapid onset of action and additional potential beneficial anti-inflammatory effects in patients with AIS. The international stroke study showed that acute treatment of stroke patients with 500mg of aspirin is safe and feasible and results in better outcome. Furthermore, the drug was safe in these circumstances with an ICH rate of only .

Therefore, the purpose of this clinical trial is to examine the safety and efficacy of the combination of aspirin with rt-TPA in patients with AIS.

DETAILED DESCRIPTION:
Background and Objectives:

Management of acute ischemic stroke consists of thrombolytic drugs aiming at opening occluded vessels. Tissue plasminogen activator (TPA) is the only drug approved by the FDA (1, 2). The use of TPA is significantly limited by a relatively narrow therapeutic window of up to 3-4.5 hours following stroke onset (3, 4). Use of TPA outside of this time window is associated with an unacceptably high risk of hemorrhage including symptomatic intracranial hemorrhage (sICH) (5, 6). While TPA is efficacious in reducing stroke associated disability its effects are limited by the phenomenon of early re-occlusion after successful reperfusion of the occluded artery.

Previous reports have shown that among patients receiving IV TPA within 3 hours of stroke onset 61% re-perfuse at 1 hour, with about 67% of these having partial recanalization and 33% complete recanalization of the occluded artery (7). reperfusion rates at 2 hours tend to be much lower ranging around 30-40% implying early re-occlusion (8). Indeed it was found that 25% of the patients that have successfully reperfused will re-occlude the artery within 2 hours (7). Re-occlusion of an already reperfused artery was more common in elderly patients with severe ipsilateral carotid stenosis and higher NIHSS scores and was associated with poor outcome (7). We speculate that re-occlusion is much more common in atherothrombotic strokes compared with embolic stroke. In embolic stroke TPA disintegrates the occluding embolus frequently and there is no remaining exposed endothelium or plaque that would trigger thrombosis (9). In contrast, in atherothrombotic stroke TPA disintegrates the occluding thrombus leading to re-perfusion less frequently (9) and the exposed thrombogenic elements within the ruptured plaque remain in place triggering repeated platelet activation and re-thrombosis.

Because primary reperfusion is less frequent in patients with atherothrombotic large vessel stroke and re-occlusion is more common in these patients and both these processes involve platelet aggregation and activation at the site of thrombosis we argue that addition of anti-platelet agent would be able to increase reperfusion rates and decrease re-occlusion rates in these patients.

Aspirin is the most commonly used antiplatelet agent in stroke patients. It has a relatively long half life and a relatively rapid onset of therapeutic effect(10, 11). Furthermore, an additional aspirin bolus may reverse a state of aspirin resistance in patients suffering a stroke while on aspirin(12, 13). Aspirin is safe when given to patients with acute stroke as soon as the diagnosis is made (14, 15).

Because the FDA approval of TPA use for stroke patients had a pre-requisite of not using concurrent anti-thrombotic drugs in the 24 hours after TPA administration the safety of aspirin needs to be studied in a randomized trial. However, it should be noted that pre-TPA aspirin use was not associated with an increased ICH risk in patients given the drug (16) and therefore pre-morbid aspirin use is not considered a contraindication for TPA administration in acute stroke.

The study will be a randomized double blind study exploring the safety of adding 500 mg of aspirin given P.O. to standard doses of IV TPA.

STUDY ENDPOINTS:

PRIMARY ENDPOINT

1. Safety (mortality, symptomatic ICH, asymptomatic ICH). SECONDARY ENDPOINTS

1. Proportion of patients achieving excellent functional outcome as determined by a modified Rankin score (mRS) < 2 and Barthel index (BI) > 85 obtained at 3 months after stroke onset.
2. Good neurological outcome as assessed by NIH stroke scale score at discharge < 5 or showing improvement of at least 8 points from the initial stroke score.
3. Good neurological outcome as assessed by NIH stroke scale score at 3 months < 5 or showing improvement of at least 8 points from the initial stroke score.

Inclusion and Exclusion Criteria

INCLUSION CRITERIA:

Patients must meet all of the inclusion criteria.

1. Diagnosis of acute ischemic stroke with onset less than 4.5 hours prior to the planned start of intravenous alteplase. Acute ischemic stroke is defined as a measurable neurological deficit of sudden onset, presumed secondary to focal cerebral ischemia. Stroke onset will be defined as the time the patient was last known to be without the new clinical deficit. Patients whose deficits have worsened in the last 4.5 hours are not eligible if their first symptoms started more than 4.5 hours before. If the stroke started during sleep, stroke onset will be recorded as the time the patient was last known to be at baseline.
2. Disabling neurological deficit attributable to acute ischemic stroke in the middle cerebral artery territory.
3. NIHSS less than or equal to 18 for left hemisphere strokes, NIHSS less than or equal to 16 for others.
4. Evidence of MCA occlusion (stem or branch) prior to drug administration by TCD, CTA or MRA.
5. Age 18-85 years, inclusive.
6. Able to sign informed consent.

EXCLUSION CRITERIA:

Patients will be excluded from study participation for any of the following reasons:

1. Current participation in another study with an investigational drug or device within, prior participation in the present study, or planned participation in another therapeutic trial, prior to the final (day 30) assessment in this trial.
2. Absence of acoustic window to insonate the MCA on the involved side.
3. Time interval since stroke onset of less than 3 hours is impossible to determine with high degree of confidence.
4. Symptoms suggestive of subarachnoid hemorrhage, even if CT or MRI scan is negative for hemorrhage.
5. Evidence of acute myocardial infarction defined as having at least two of the following three features: 1) Chest pain suggestive of cardiac ischemia; 2) EKG findings of ST elevation of more greater than 0.2 mV in 2 contiguous leads, new onset left bundle branch block, ST segment depression, or T-wave inversion; 3) Elevated troponin I.
6. Acute Pericarditis.
7. Women known to be pregnant, lactating or having a positive or indeterminate pregnancy test.
8. Neurological deficit that has led to stupor or coma (NIHSS level of consciousness [item I a] score greater than or equal to 2).
9. High clinical suspicion of septic embolus.
10. Minor stroke with non-disabling deficit or rapidly improving neurological symptoms.
11. Baseline NIHSS greater than 18 for left hemisphere stroke or greater than 16 for others.
12. Evidence of acute or chronic ICH by head CT or MRI.
13. CT or MRI evidence of non-vascular cause for the neurological symptoms.
14. Signs of mass effect causing shift of midline structures on CT or MRI.
15. Persistent hypertension with systolic BP greater than 185 mmHg or diastolic BP greater than 110 mmHg (mean of 3 consecutive arm cuff readings over 20-30 minutes), not controlled by antihypertensive therapy or requiring nitroprusside for control.
16. Anticipated need for major surgery within 72 hours after start of study drugs, e.g., carotid endarterectomy, hip fracture repair.
17. Any intracranial surgery, intraspinal surgery, or serious head trauma (any head injury that required hospitalization) within the past 3 months.
18. Stroke within the past 3 months.
19. History of ICH at any time in the past.
20. Major trauma at the time of stroke, e.g., hip fracture.
21. Blood glucose greater than 200 mg/dl.
22. Presence or history of intracranial neoplasm (except small meninigiomas) or arteriovenous malformation.
23. Intracranial aneurysm, unless surgically or endovascularly treated more than 3 months before.
24. Seizure at the onset of stroke.
25. Active internal bleeding.
26. Major hemorrhage (requiring transfusion, surgery or hospitalization) in the past 21 days.
27. Major surgery, serious trauma, lumbar puncture, arterial puncture at a non-compressible site, or biopsy of a parenchymal organ in last 14 days. Major surgical procedures include but are not limited to the following: major thoracic or abdominopelvic surgery, neurosurgery, major limb surgery, carotid endarterectomy or other vascular surgery, and organ transplantation. For non-listed procedures, the operating surgeon should be consulted to assess the risk.
28. Presumed or documented history of vasculitis.
29. Known systemic bleeding or platelet disorder, e.g., von Willebrand's disease, hemophilia, ITP, TTP, others.
30. Platelet counts less than 100,000 cells/micro L.
31. Congenital or acquired coagulopathy (e.g., secondary to anticoagulants) causing either of the following:

    1. Activated partial thromboplastin time (aPTT) prolongation greater than 2 seconds above the upper limit of normal for local laboratory, except if due to isolated factor XII deficiency.
    2. INR greater than or equal to 1.4. Patients receiving warfarin prior to entry are eligible provided INR is less than 1.4 and warfarin can be safely discontinued for at least 48 hours.
32. Life expectancy less than 3 months.
33. Other serious illness, e.g., severe hepatic, cardiac, or renal failure; acute myocardial infarction; or complex disease that may confound treatment assessment.
34. Severe renal failure: Serum creatinine greater than 4.0 mg/dL or dependency on renal dialysis.
35. AST or ALT greater than 3 times the upper limit of normal for the local laboratory.
36. Treatment of the qualifying stroke with any thrombolytic, anti-thrombotic or GPIIbIIIa inhibitor outside of this protocol.
37. Any administration of a thrombolytic drug in the prior 7 days.
38. Treatment of the qualifying stroke with intravenous heparin unless aPTT prolongation is no greater than 2 seconds above the upper limit of normal for local laboratory prior to study drug initiation.
39. Treatment of the qualifying stroke with a low molecular weight heparin or heparinoid.
40. Known hypersensitivity to TPA.
41. Anticoagulation (evidenced by abnormal INR, aPTT, or platelet count) caused by herbal therapy.

METHOD:

Eligible patients (n=20/group) will be recruited after obtaining informed consent. Patients will be randomized to receive rt-TPA 0.9mg/kg (10% of the total dose as an IV bolus and the reminder IV over 60 minutes) + placebo or rt-TPA 0.9mg/kg + aspirin P.O. at a dose of 500mg at the time of TPA administration.. Randomization will be accomplished using an IVRS automated system. Randomization will be into time tiers of 0-1.5 hours from symptom onset, 1.5-3 hours from symptom onset and 3-4.5 hours from symptom onset for each dose tier. Overall 60 patients (30 TPA + active drug and 30 TPA only are to be recruited). Study medications will be supplied by the hospital and will have a total volume, color and odor that will be identical to placebo. At the end of recruitment the randomization codes will be opened and the data safety monitoring board (DSMB) will determine the safety of continuing the study in the next dose tier. Samples will be collected for safety data (renal, hepatic and coagulation studies) and sent to local laboratories in each center. Investigators will be notified immediately on any lab results by fax and email. ECGs will be read at a central facility and investigators will be notified on any abnormal result immediately via fax and email. All AE and SAE will be reported immediately.

EVALUATIONS

Safety:

Hemodynamics: Patients will be monitored non-invasively for blood pressure, heart rate, oxygen saturation q2rhs in the first 24 hours post stroke and then every 6 hours for the next 24 hours and then every 12 hours for the reminder of the hospitalization.

Coagulation tests: PT, PTT and PLT blood counts will be evaluated daily in the first 3 days of hospitalization.

Blood tests: Blood chemistry, liver function tests and cardiac enzymes will be evaluated daily for the first 3 days and then at discharge.

Cardiac rhythm: ECG will be evaluated daily on a 12 lead recording on the first 3 days of hospitalization and then at discharge.

CT: Brain CT will be obtained prior to drug administration and in included patients repeated scans will be obtained at 96-120 hours to evaluate final infarct size. In cases of suspected hematoma brain CT would be obtained immediately and the number of patients sustaining an ICH following drug administration will be recorded.

All other adverse events (AE) and serious adverse events (SAE) will be recorded and promptly evaluated by the data safety monitoring board that will decide whether or not these events are drug related and which will have the authority to prematurely terminate the study in case an unexpected SAE emerges and appears to be drug related. AE and SAE will be defined conventionally such that AE is any adverse event and SAE as an AE necessitating prolongation of hospitalization or any adverse event that is potentially life threatening).

NEUROLOGICAL Included patients will be examined before and after randomization with the National Institute of Health stroke scale (NIHSS) on days 1,2,3,5 and discharge and on outpatient visits at months 1 and 3-post stroke.

FUNCTIONAL OUTCOME Patients will be evaluated with the Barthel index (BI) and modified Rankin score (MRS) administered on discharge day and during outpatient visits at month 1 and 3-post stroke.

References:

1. Tissue plasminogen activator for acute ischemic stroke. The National Institute of Neurological Disorders and Stroke rt-PA Stroke Study Group. N Engl J Med. 1995;333:1581-1587
2. Hacke W, Kaste M, Fieschi C et al. Intravenous thrombolysis with recombinant tissue plasminogen activator for acute hemispheric stroke. The European Cooperative Acute Stroke Study (ECASS). JAMA. 1995;274:1017-1025
3. Albers GW, Bates VE, Clark WM et al. Intravenous tissue-type plasminogen activator for treatment of acute stroke: the Standard Treatment with Alteplase to Reverse Stroke (STARS) study. JAMA. 2000;283:1145-1150
4. Hacke W, Donnan G, Fieschi C et al. Association of outcome with early stroke treatment: pooled analysis of ATLANTIS, ECASS, and NINDS rt-PA stroke trials. Lancet. 2004;363:768-774
5. Graham GD. Tissue plasminogen activator for acute ischemic stroke in clinical practice: a meta-analysis of safety data. Stroke. 2003;34:2847-2850
6. Burgin WS, Staub L, Chan W et al. Acute stroke care in non-urban emergency departments. Neurology. 2001;57:2006-2012
7. Rubiera M, Alvarez-Sabin J, Ribo M et al. Predictors of early arterial reocclusion after tissue plasminogen activator-induced recanalization in acute ischemic stroke. Stroke. 2005;36:1452-1456
8. Molina CA, Ribo M, Rubiera M et al. Microbubble administration accelerates clot lysis during continuous 2-MHz ultrasound monitoring in stroke patients treated with intravenous tissue plasminogen activator. Stroke. 2006;37:425-429
9. Molina CA, Montaner J, Arenillas JF et al. Differential pattern of tissue plasminogen activator-induced proximal middle cerebral artery recanalization among stroke subtypes. Stroke. 2004;35:486-490
10. Barnett HJ. Aspirin in stroke prevention. An overview. Stroke. 1990;21:IV40-43
11. Schror K. Antiplatelet drugs. A comparative review. Drugs. 1995;50:7-28
12. Wang TH, Bhatt DL, Topol EJ. Aspirin and clopidogrel resistance: an emerging clinical entity. Eur Heart J. 2006;27:647-654
13. Sztriha LK, Sas K, Vecsei L. Aspirin resistance in stroke: 2004. J Neurol Sci. 2005;229-230:163-169
14. The International Stroke Trial (IST): a randomised trial of aspirin, subcutaneous heparin, both, or neither among 19435 patients with acute ischaemic stroke. International Stroke Trial Collaborative Group. Lancet. 1997;349:1569-1581
15. CAST: randomised placebo-controlled trial of early aspirin use in 20,000 patients with acute ischaemic stroke. CAST (Chinese Acute Stroke Trial) Collaborative Group. Lancet. 1997;349:1641-1649
16. Levy DE, Brott TG, Haley EC, Jr. et al. Factors related to intracranial hematoma formation in patients receiving tissue-type plasminogen activator for acute ischemic stroke. Stroke. 1994;25:291-297

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the inclusion criteria.

1. Diagnosis of acute ischemic stroke with onset less than 4.5 hours prior to the planned start of intravenous alteplase. Acute ischemic stroke is defined as a measurable neurological deficit of sudden onset, presumed secondary to focal cerebral ischemia. Stroke onset will be defined as the time the patient was last known to be without the new clinical deficit. Patients whose deficits have worsened in the last 4.5 hours are not eligible if their first symptoms started more than 4.5 hours before. If the stroke started during sleep, stroke onset will be recorded as the time the patient was last known to be at baseline.
2. Disabling neurological deficit attributable to acute ischemic stroke in the middle cerebral artery territory.
3. NIHSS less than or equal to 18 for left hemisphere strokes, NIHSS less than or equal to 16 for others.
4. Evidence of MCA occlusion (stem or branch) prior to drug administration by TCD, CTA or MRA.
5. Age 18-85 years, inclusive.
6. Able to sign informed consent.

   For MRI Arm only:
7. Screening MRI diagnostic of focal cerebral ischemia corresponding to the clinical deficits. The MRI evaluation must involve echo planar diffusion weighted imaging, MRA, and MRI perfusion. A normal appearing MRA with an appropriate perfusion deficit is eligible. An apparent stenosis or occlusion on MRA with normal appearing perfusion distally will not be eligible. Poor quality or uninterpretable MRA will not make patient ineligible. Patients who have a normal appearing DWI are eligible.
8. Evidence on PWI MRI or a perfusion defect corresponding to the acute stroke syndrome. The PWI will be assessed by relative mean transit time (MTT) images obtained prior to the start of rt-TPA therapy.

Exclusion Criteria:

Patients will be excluded from study participation for any of the following reasons:

1. Current participation in another study with an investigational drug or device within, prior participation in the present study, or planned participation in another therapeutic trial, prior to the final (day 30) assessment in this trial.
2. Absence of acoustic window to insonate the MCA on the involved side.
3. Time interval since stroke onset of less than 3 hours is impossible to determine with high degree of confidence.
4. Symptoms suggestive of subarachnoid hemorrhage, even if CT or MRI scan is negative for hemorrhage.
5. Evidence of acute myocardial infarction defined as having at least two of the following three features: 1) Chest pain suggestive of cardiac ischemia; 2) EKG findings of ST elevation of more greater than 0.2 mV in 2 contiguous leads, new onset left bundle branch block, ST segment depression, or T-wave inversion; 3) Elevated troponin I.
6. Acute Pericarditis.
7. Women known to be pregnant, lactating or having a positive or indeterminate pregnancy test.
8. Neurological deficit that has led to stupor or coma (NIHSS level of consciousness [item I a] score greater than or equal to 2).
9. High clinical suspicion of septic embolus.
10. Minor stroke with non-disabling deficit or rapidly improving neurological symptoms.
11. Baseline NIHSS greater than 18 for left hemisphere stroke or greater than 16 for others.
12. Evidence of acute or chronic ICH by head CT or MRI.
13. CT or MRI evidence of non-vascular cause for the neurological symptoms.
14. Signs of mass effect causing shift of midline structures on CT or MRI.
15. Persistent hypertension with systolic BP greater than 185 mmHg or diastolic BP greater than 110 mmHg (mean of 3 consecutive arm cuff readings over 20-30 minutes), not controlled by antihypertensive therapy or requiring nitroprusside for control.
16. Anticipated need for major surgery within 72 hours after start of study drugs, e.g., carotid endarterectomy, hip fracture repair.
17. Any intracranial surgery, intraspinal surgery, or serious head trauma (any head injury that required hospitalization) within the past 3 months.
18. Stroke within the past 3 months.
19. History of ICH at any time in the past.
20. Major trauma at the time of stroke, e.g., hip fracture.
21. Blood glucose greater than 200 mg/dl.
22. Presence or history of intracranial neoplasm (except small meninigiomas) or arteriovenous malformation.
23. Intracranial aneurysm, unless surgically or endovascularly treated more than 3 months before.
24. Seizure at the onset of stroke.
25. Active internal bleeding.
26. Major hemorrhage (requiring transfusion, surgery or hospitalization) in the past 21 days.
27. Major surgery, serious trauma, lumbar puncture, arterial puncture at a non-compressible site, or biopsy of a parenchymal organ in last 14 days. Major surgical procedures include but are not limited to the following: major thoracic or abdominopelvic surgery, neurosurgery, major limb surgery, carotid endarterectomy or other vascular surgery, and organ transplantation. For non-listed procedures, the operating surgeon should be consulted to assess the risk.
28. Presumed or documented history of vasculitis.
29. Known systemic bleeding or platelet disorder, e.g., von Willebrand's disease, hemophilia, ITP, TTP, others.
30. Platelet counts less than 100,000 cells/micro L.
31. Congenital or acquired coagulopathy (e.g., secondary to anticoagulants) causing either of the following:

    1. Activated partial thromboplastin time (aPTT) prolongation greater than 2 seconds above the upper limit of normal for local laboratory, except if due to isolated factor XII deficiency.
    2. INR greater than or equal to 1.4. Patients receiving warfarin prior to entry are eligible provided INR is less than 1.4 and warfarin can be safely discontinued for at least 48 hours.
32. Life expectancy less than 3 months.
33. Other serious illness, e.g., severe hepatic, cardiac, or renal failure; acute myocardial infarction; or complex disease that may confound treatment assessment.
34. Severe renal failure: Serum creatinine greater than 4.0 mg/dL or dependency on renal dialysis.
35. AST or ALT greater than 3 times the upper limit of normal for the local laboratory.
36. Treatment of the qualifying stroke with any thrombolytic, anti-thrombotic or GPIIbIIIa inhibitor outside of this protocol.
37. Any administration of a thrombolytic drug in the prior 7 days.
38. Treatment of the qualifying stroke with intravenous heparin unless aPTT prolongation is no greater than 2 seconds above the upper limit of normal for local laboratory prior to study drug initiation.
39. Treatment of the qualifying stroke with a low molecular weight heparin or heparinoid.
40. Known hypersensitivity to TPA.
41. Anticoagulation (evidenced by abnormal INR, aPTT, or platelet count) caused by herbal therapy.

    FOR non-MRI arm only (#42-43):
42. Ischemic changes on screening CT of greater than approximately one third of the territory of the middle cerebral artery territory by qualitative assessment.
43. Patients who were excluded by screening MRI, except for exclusions #45 (contraindication to MRI) and #46 (PWI was not obtained or is uninterpretable) and #50 (MRI not obtainable because it would have put the patient out of the 3 hour time window for alteplase).

    FOR MRI arm only (#44-51):
44. Contraindication to MRI scan.
45. PWI not obtained or uninterpretable.
46. No MTT defect corresponding to acute stroke deficit.
47. DWI abnormality larger than approximately one third of the territory of the middle cerebral artery territory by qualitative assessment.
48. Satellite DWI hyperintensity with corresponding hyperintensity on T2 weighted image or FLAIR in a vascular territory different than the index stroke (this is evidence of a new ischemic lesion greater than 3 hours in duration).
49. Evidence of multiple microbleeds on gradient echo MRI (GRE).
50. MRI not obtained because it would have put the patient out of the 3 hour time window for alteplase.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-03; Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
PRIMARY ENDPOINT
Safety (mortality, symptomatic ICH, asymptomatic ICH).

SECONDARY OUTCOMES:
Proportion of patients achieving excellent functional outcome as determined by a modified Rankin score (mRS) < 2 and Barthel index (BI) > 85 obtained at 3 months after stroke onset.
Good neurological outcome as assessed by NIH stroke scale score at discharge < 5 or showing improvement of at least 8 points from the initial stroke score.
Good neurological outcome as assessed by NIH stroke scale score at 3 months < 5 or showing improvement of at least 8 points from the initial stroke score.

CONTACTS AND LOCATIONS:
Overall Officials: Ronen R Leker, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah University Medical Center, Jerusalem, Israel